CLINICAL TRIAL: NCT06138587
Title: Cytokine-induced Memory-like Natural Killer Cell Therapy After Hematopoietic Stem Cell Transplantation for Eradication of Measurable Residual Disease, a Phase I/Ib Clinical Trial
Brief Title: Preemptive CIML NK Cell Therapy After Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Roman Shapiro, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-535
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Leukemia; Leukemia, Myeloid; Myelodysplastic Syndromes; Myeloproliferative Neoplasm; Myeloproliferative Disorders
Keywords: Acute Myeloid Leukemia; Leukemia; Leukemia, Myeloid; Myelodysplastic Syndrome; MDS and Myeloproliferative Neoplasm Overlap Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Leukemia, Myeloid; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1/1b: CIML NK Cells + Interleukin-2 (Experimental): 5 eligible participants will be enrolled to determine the maximum tolerated dose (MTD) of CIML NK at starting dose level 0.
  * Screening and baseline visit with assessments and bone marrow aspirate and biopsy.
  * Day 0: Standard-of-care conditioning chemotherapy and stem cell infusion.
  * Day 7: Predetermined dose of CIML NK cells 1x daily.
  * Days 7, 9, 11, 13, 15: Predetermined dose of Interleukin-2 1x daily every other day (5 doses total).
  * Dose limiting toxicity period for 6 weeks after infusion of CIML NK cells
  If 0 or 1 dose limiting toxicity is observed at the dose level, then this dose will be the MTD and study will proceed to Phase 1b.
  De-escalation to dose level -1 per protocol if ≥2 DLTs occur with dose Level 0.
  In phase Ib, 10 additional participants will be enrolled at the maximum tolerated dose.
  Interventions: Biological: Cytokine Induced Memory-like Natural Killer Cells; Biological: Interleukin-2

INTERVENTIONS:
Biological: Cytokine Induced Memory-like Natural Killer Cells — Allogeneic, cytokine induced memory-like natural killer cells, via intravenous infusion per protocol.
  Other Names: CIML NK cells
Biological: Interleukin-2 — Recombinant, human glycoprotein, single-use 22 MIU vials, via subcutaneous injection per protocol.
  Other Names: Aldesleukin, Proleukin

SUMMARY:
The purpose of this research study is to test the safety and efficacy of cytokine induced memory-like (CIML) natural killer (NK) cells expanded with Interleukin-2 (IL-2) at preventing relapse in acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), or MDS and myeloproliferative neoplasm (MPN) overlap syndrome after a standard-of-care stem cell transplant.

Names of the study therapies involved in this study are:

* CIML NK cells intravenous infusion (cellular therapy)
* Subcutaneous Interleukin-2 (recombinant, human glycoprotein)

DETAILED DESCRIPTION:
This is a phase I/Ib study of the pre-emptive treatment using related donor-derived cytokine induced memory-like (CIML) natural killer (NK) cells combined with Interleukin-2 (IL-2) for participants with acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), and MDS/myeloproliferative neoplasm (MDS/MPN) overlap syndrome at high risk for post-allogeneic stem cell transplant (SCT) relapse.

The U.S. Food and Drug Administration (FDA) has not approved CIML NK cells as a treatment for AML, MDS or MDS and MPN overlap syndrome.

The research study procedures include screening for eligibility, intravenous infusion of CIML NK cells in the hospital, standard-of-care stem cell infusion, subcutaneous interleukin-2 (IL-2) infusions, x-rays, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, Positron Emission Tomography (PET) scans, blood tests, bone marrow biopsies, echocardiograms, and electrocardiograms.

Participation in this research study is expected to last up to 3 years.

It is expected that up to 30 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria for Trial Enrollment:

* Histologically or cytologically confirmed diagnosis of AML, MDS, or MDS/MPN that is at high risk for post-transplant relapse and that has measurable disease prior to transplant, except for patients with TP 53 mutated disease who are eligible regardless of measurable residual disease. Patients at high risk for post-transplant relapse include:

  * De novo AML diagnosed at or after age 60, except CBF AML
  * De novo AML in CR1 AND MRD+ by Hematologics Inc. flow cytometry pretransplant (this would be on the most recent pre-transplant bone marrow)
  * Secondary AML
  * Any AML transplanted in CR2 or greater
  * TP53-mutated MDS or AML
  * Therapy-related MDS or AML
  * MDS with monosomy 7
  * MDS with >= 10% blasts at the time of transplant
  * MDS/MPN or CMML
* Adequate organ function within 2 weeks of NK cell infusion as defined below (should correspond with admission for SCT):

  * Total bilirubin: ≤1.5 x institutional upper limit of normal (ULN) (except Gilbert's or disease related hemolysis, then < 3 x ULN)
  * AST(SGOT)/ALT(SGPT): ≤3 x institutional ULN
  * Serum creatinine </= 2.0mg/dL
  * O2 saturation: ≥90% on room air
  * LVEF >40%. If there is no clinical evidence of a change in cardiovascular function from the time of pre-transplantation ECHO (per FACT standards should be performed within 6 weeks of stem cell infusion), then there is no need to repeat it. Otherwise, an ECHO will need to be repeated.
* Adult patients (age ≥ 18) eligible for and planned to undergo a standard-of-care reduced intensity conditioning (RIC) HLA-matched related or related haploidentical allogeneic stem cell transplant using PTCY-based GVHD prophylaxis. All eligibility criteria and workups for undergoing SOC allogeneic SCT for the recipient and donor will be based on institutional standards and SOPs.
* For patients with AML, the disease must meet criteria for CR/Cri according to 2017 ELN guidelines. For patients with MDS and MDS/MPN patients, the blast percentage on the bone marrow aspirate and biopsy must be less than 10%.
* The same related donor is available to provide a non-mobilized apheresis product after the stem-cell donation.
* ECOG performance status <= 2 (Karnofsky >= 60%, see Appendix C).
* Negative pregnancy test for women of childbearing age
* The effects of CIML NK cells combined with IL-2 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after IL-2 dose administration.
* No laboratory evidence of ongoing hemolysis in opinion of investigator

Exclusion Criteria Trial Enrollment:

* Adult participants who are eligible for and who would be expected to have a greater benefit from myeloablative conditioning in their SOC allo HSCT as judged by their treating physician
* Participants with mutations such as FLT3-ITD, IDH, or BCR-ABL mutations who are planned to receive targeted agent maintenance therapy to prevent relapse post-transplant are excluded.
* Extramedullary leukemia involving sanctuary sites not readily accessible to immune surveillance, such as CNS or testis. Other sites of extramedullary relapse (e.g., leukemia cutis, granulocytic sarcoma) are acceptable.
* The planned use of sirolimus for GVHD prophylaxis would result in exclusion of the patient from the study. Consideration of the addition of sirolimus to the GVHD prophylaxis regimen within the first 100 days after transplant must be reviewed with the study PI.
* Prior history of allogeneic stem cell transplant other than SOC alloHSCT referred to in this study taking place 7 days prior to CIML NK infusion.
* Prior history of solid organ (allograft) transplantation
* Prior history of allergic reactions to cellular products
* Uncontrolled concurrent illness such as ongoing or active infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, or psychiatric/social illness that would limit compliance with study requirements.
* Pregnant women are excluded from this study because of the unknown teratogenic risk of CIML NK cells and IL-2 and with the potential for teratogenic or abortifacient effects by Flu/Cy chemotherapy regimen. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CIML NK cells and IL-2, breastfeeding should be discontinued if the mother is treated on this study.
* HIV-positive patients are excluded due to the potential for interaction between antiretroviral therapy as well as the risk for lethal infection in the context of marrow-suppressive therapy.
* Patients with active and uncontrolled Hepatitis B or C are ineligible due to the high risk of treatment-related hepatotoxicity after cellular therapy.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: 1. History of other malignancy and have had complete remission of disease for at least 2 years; 2. Diagnosed and treated within the past 2 years for: nonmetastatic melanoma, surgically resected (not needing systemic chemotherapy) squamous cell carcinoma of skin and nonmetastatic prostate cancer not needing systemic chemotherapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to IL-2 or other agents used in study. 3. Diagnosed with MGUS or smoldering myeloma, and/or treated for multiple myeloma or plasmacytoma as long as attainment of complete remission by IMWG criteria following therapy.
* Prior history of Grade 2 or higher hemolytic anemia (>/= 2g decrease in hemoglobin plus laboratory evidence of hemolysis) from any cause.

Inclusion Criteria to Receive CIML NK Infusion

* Adequate organ function within 24 hours of NK cell infusion as defined below:

  * Total bilirubin: ≤1.5 x institutional upper limit of normal (ULN) (except Gilbert's or disease-related hemolysis, then < 3 x ULN)
  * AST(SGOT)/ALT(SGPT): ≤3 x institutional ULN
  * Grade ≥3 non-hematologic toxicities of cyclophosphamide and fludarabine conditioning (except for Grade 3 nausea, vomiting, diarrhea, or constipation).
* No significant change in clinical status that would, in the opinion of the investigator, increase the risk of adverse events associated with CIML NK infusion, (e.g., symptomatic congestive heart failure, unstable angina, cardiac arrhythmia)
* No evidence of ongoing hemolysis in opinion of investigator

Exclusion Criteria to Receive CIML NK Infusion:

* Systemic steroid therapy (oral or IV) on the day of NK cell infusion
* Uncontrolled concurrent illness such as ongoing or active infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, or psychiatric/social illness that would limit compliance with study requirements.
* Participants who have had other investigational agents within 4 weeks prior to CIML NK cell infusion (6 weeks for nitrosoureas or mitomycin C), or immunotherapy within 8 weeks prior, or those who have not recovered from adverse events due to agents administered more than 4 weeks prior. Therapy with BCR-ABL inhibitors must be stopped at least 2 weeks before CIML NK cell infusion and may not be resumed during the DLT period. The use of tocilizumab for cytokine release syndrome after stem cell infusion does not exclude patients, but the use of steroids for the treatment of CRS excludes patients if they are still on steroids by the day of planned NK cell infusion.
* Systemic steroid use of >10mg/day of prednisone equivalent is an exclusion criteria unless there is a plan for dose to be tapered below this limit within 4 weeks prior to NK cell infusion.

Patients must be off systemic steroid therapy on the day of planned NK cell infusion.

-The presence of donor-specific antibodies (DSAs) with mean fluorescence intensity (MFI) >1000 using a standard assay who do not receive a desensitization protocol prior to and during stem cell transplant, or else who do receive a desensitization protocol and have detectable DSAs +1 day after stem cell infusion.

If inclusion/exclusion criteria are not met on planned day of CIML NK cell infusion, the NK cell infusion may be delayed for up to 48 hours to enable inclusion criteria to be met.

However, patient may still receive CIML NK infusion if relevant parameters are reviewed and both PI and IND holder are in agreement with proceeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) [Phase 1] | 6 weeks
  All DLT was defined as an adverse event (AE) that is related to the CIML NK cell infusion combined with IL-2 in adult patients undergoing RIC HLA-matched related or haploidentical donor stem cell transplantation using PTCY-based GVHD prophylaxis. Toxicities are to be assessed according to the CTCAEv5 (Appendix C). Management and dose modifications associated with the above adverse events are outlined in protocol 6.

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) [Phase 1] | 6 weeks
  The MTD in the CIML NK cell infusion combined with IL-2 in adult patients undergoing RIC HLA-matched related or haploidentical donor stem cell transplantation using PTCY-based GVHD prophylaxis is determined by the number pf patients who experience a DLT. See previous primary outcome measure for the DLT definition. The MTD is defined as the highest dose at which fewer than 2 out of 5 patient in each dose cohort experience a DLT. Dose-de-escalation will take place if MTD considered exceeded in each dose cohort.
Complete Remission (CR/CRi) Rate (CRR) | 100 days
  The CRR is defined as the proportion of participants achieving complete remission (CR) or complete remission with incomplete hematologic recovery (CRi) based on criteria defined in protocol appendix H.
Measurable Residual Disease (MRD) Rate | At 35 and 100 days
  MRD rate is defined as the proportion pf participants achieving MRD using the validated NGS-based assay.
1-year Progression-Free Survival (PFS) Rate | 1 year
  1-year PFS is a probability estimated using progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) or death, or is censored at time of last disease assessment.
1-year Overall Survival (OS) | 1 year
  1-year OS is a probability estimated using the Kaplan-Meier method; OS is defined as the time from study entry to death, or censored at date last known alive.
6-month Graft-versus-host Disease (GVHD) and Relapse Free Survival (GRFS) | 6 months
  6-month GRFS is a probability estimated using the Kaplan-Meier method. GVHD-free relapse-free survival (GRFS) is defined as grade 3-4 acute GVHD, chronic GVHD requiring systemic treatment, relapse, or death. GVHD assessment detail in protocol appendix G.
12-month Graft-versus-host Disease (GVHD) and Relapse Free Survival (GRFS) | 12 months
  12-month GRFS is a probability estimated using the Kaplan-Meier method. GVHD-free relapse-free survival (GRFS) is defined as grade 3-4 acute GVHD, chronic GVHD requiring systemic treatment, relapse, or death. GVHD assessment detail in protocol appendix G.
100-day Acute GVHD Rates | 100 days
  Acute GVHD will be estimated in the competing risks framework treating death or relapse without developing GVHD as a competing event. GVHD assessment detail in protocol appendix G.
6-month Acute GVHD Rates | 6 months
  Acute GVHD will be estimated in the competing risks framework treating death or relapse without developing GVHD as a competing event. GVHD assessment detail in protocol appendix G.
12-month Chronic GVHD Rates | 12 months
  Chronic GVHD will be estimated in the competing risks framework treating death or relapse without developing GVHD as a competing event. GVHD assessment detail in protocol appendix G.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Shapiro, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu